CLINICAL TRIAL: NCT00831350
Title: Posterior Vitreous Detachment (PVD) Assessment During Dual RVO Lucentis Evaluations (PADDLE Study)
Brief Title: Posterior Vitreous Detachment (PVD) Assessment During Dual Retinal Vein Occlusion (RVO) Lucentis Evaluations
Acronym: PADDLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barnes Retina Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Rhonda Weeks, Nancy M. Holekamp, MD, Barnes Retina Institute
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4348s; 09-0049
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Retinal Vein Occlusion; Posterior Vitreous Detachment
Keywords: RVO; PVD
MeSH Terms: conditions — Retinal Vein Occlusion; Vitreous Detachment | interventions — Ranibizumab

STUDY DESIGN:
Intervention Model Description: BRVO and CRVO will be enrolled in this trial.
Oversight: Data Monitoring Committee: No

ARMS (1):
- ranibizumab (Experimental)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Subjects will receive study medication ranibizumab 0.5mg. Re-treatment will occur monthly through 6 injections
  Other Names: Lucentis

SUMMARY:
This is a study of subjects with retinal vein occlusion (RVO) specifically looking at the difference in outcomes between patients with posterior vitreous detachment (PVD) and those without PVD. Posterior vitreous detachment is a condition where the gel-like substance that occupies the space between the retina and the lens of the eye liquefies and separates from the retina. 20 subjects from Barnes Retina Institute will be enrolled in this study. Based on a pre-treatment ultrasound (a test utilizing high-frequency sound waves to look at the inside of the eye), high resolution OCT (a noninvasive procedure called optical coherence tomography to check the thickness of your retina) and clinical exam, subjects will be assigned to one of 2 groups at baseline: Group 1 will be those with PVD and Group 2 will be those without PVD. Then subjects will receive monthly intravitreal (inside the eye) injections of Ranibizumab.

DETAILED DESCRIPTION:
Several retinovascular diseases have been shown to be VEGF dependent including retinal vein occlusion, wet age-related macular degeneration, and diabetic retinopathy. The role of the vitreous or composition of the vitreous cavity has been examined in diabetic retinopathy on many occasions in the past and clinically it has been felt that a posterior vitreous separation leads a quieting and involution of diabetic retinopathy, both proliferative as well as pre-proliferative retinopathy. This clinical observation has never had any basic science data to support it. However, it has recently been shown that in cat eyes with posterior vitreous separation the vitreous cavity has a much lower VEGF concentration than in cat eyes with an attached posterior vitreous. This may be due to the fact that flow of oxygen from the retinal vasculature is increased by PVD. Vitreous oxygen levels are inversely associated with vitreous VEGF levels. As oxygen tension increases, VEGF levels will decline. This suggests if higher amounts of VEGF are present in the eye without PVD perhaps a powerful anti-VEGF drug, such as ranibizumab, may be of greater benefit to treat VEGF dependent retinovascular disease. To try and answer this question clinically, we have suggested that an analysis of the vitreous status in treatment naive eyes with retinal vein occlusion beginning ranibizumab therapy be undertaken to see if eyes without a posterior vitreous separation would achieve greater improvement in vision and a return to more normal retinal physiology compared to eyes with a posterior vitreous separation. No study has assessed PVDs in RVO patients receiving potential treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Subjects of either gender, Age > 18 years
* Best corrected visual acuity in the study eye between 20/40 and 2/200 inclusive.
* Retinal venous occlusive disease (BRVO or CRVO)
* Clear ocular media and adequate papillary dilation to permit good quality stereoscopic fundus photography, scheimpflug photography and high resolution OCT
* Ability to return for all study visits

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation.
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Prior RVO in the study eye
* Duration of RVO greater than 6 months
* Laser photocoagulation for macular edema within 3 months of Day 0
* Patients prior eye treatment including anti-VEGF therapy (within 3 months) or, intravitreal corticosteroid therapy (within 6 months)
* Prior vitreoretinal surgery.
* Had ocular surgery within the past 60 days in the study eye.
* Concurrent use of more than two therapies for glaucoma.
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure >30 mm Hg despite treatment with anti-glaucoma medication).
* Neovascular glaucoma
* Concurrent use of systemic anti-VEGF agents
* Has active infection in the study eye.
* Inability to obtain photographs.
* Has received investigational therapy within 60 days prior to study entry.
* Patients with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
* Has other conditions the investigator considers to be sound reasons for exclusion (e.g., lack of motivation, history of poor compliance, concomitant illnesses, personality disorder, mental condition, drug abuse, use of neuroleptics, physical or social condition predicting difficulty in long-term follow-up).
* Has an allergy to fluorescein sodium dye.
* Inability to comply with study or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mean change in BCVA at 6 months in the PVD positive and PVD negative ranibizumab-treated groups. | 6 months

SECONDARY OUTCOMES:
To measure the mean change in central retinal thickness per OCT from baseline to Month 6 in PVD (+) and PVD (-) patients. | 6 months
To measure the mean change in leakage as determined by FA from baseline to Month 6 in PVD (+) and PVD (-) patients. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Holekamp, MD, Principal Investigator — Barnes Retina Institute
Locations (1):
- Barnes Retina Institute, St Louis, Missouri, United States